CLINICAL TRIAL: NCT03766971
Title: Influence of Tobacco Use on Cannabis Use
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: In response to quality assurance and compliance concerns, OHRP issued an FWA restriction on NYSPI research that included a pause of human research as of June 23, 2023.
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Margaret Haney, Professor of Psychiatry, Columbia University, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 7707
Record Dates: First submitted 2018-12-04; First posted 2018-12-06 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Cannabis Use; Tobacco Use
MeSH Terms: conditions — Tobacco Use | interventions — nabiximols

STUDY DESIGN:
Intervention Model Description: The effects of 7- and 21-days of tobacco cessation on cannabis relapse in daily cigarette-smoking, cannabis smokers will be compared, with half the participants in each group initiating tobacco cigarette smoking early (<16 years) and the other half later (>=16 years).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Research staff will be blind to the age of tobacco onset condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Early-onset Cigarette Smokers (Experimental): Participants who began smoking cigarettes earlier in life (<16 years old) will be randomized to 7 or 21 days of tobacco cessation.
  Interventions: Behavioral: 7 days of Tobacco Cessation; Behavioral: 21 days of Tobacco Cessation; Drug: Cannabis
- Late-onset Cigarette Smokers (Experimental): Participants who began smoking cigarettes later in life (>16 years old) will be randomized to 7 or 21 days of tobacco cessation.
  Interventions: Behavioral: 7 days of Tobacco Cessation; Behavioral: 21 days of Tobacco Cessation; Drug: Cannabis

INTERVENTIONS:
Behavioral: 7 days of Tobacco Cessation — Participants will be randomly assigned to 7 days of tobacco cessation.
  Other Names: Early onset
Behavioral: 21 days of Tobacco Cessation — Participants will be randomly assigned to 21 days of tobacco cessation.
  Other Names: Late onset
Drug: Cannabis — Participants will receive cannabis.

SUMMARY:
Cannabis smokers who also smoke tobacco cigarettes have markedly higher rates of cannabis relapse relative to those who do not use tobacco. There is a clear need to develop and evaluate interventions for dual tobacco and cannabis users. The investigators of this study have previously shown that the co-use of tobacco cigarettes contributes to the maintenance of daily cannabis use, and that age of cigarette onset is a critical predictor of treatment outcome. Short-term tobacco cessation may suffice in altering cannabis relapse rates in later-onset cigarette smokers, while a longer period of tobacco cessation may be needed for earlier-onset smokers. In the current study, a human laboratory model will be utilized to determine whether cannabis relapse varies as a function of tobacco cessation duration and age of tobacco use onset.

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant females aged 18-60 years old
* Use cannabis
* Smoke tobacco cigarettes
* Medically and psychologically healthy

Exclusion Criteria:

* Regular drug use other than cannabis
* Current pregnancy/lactation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Cannabis self-administration | During 9-day inpatient phase
  Number of cannabis cigarettes participant chooses to smoke.

CONTACTS AND LOCATIONS:
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided